CLINICAL TRIAL: NCT05084261
Title: A Multicenter, Randomized, Placebo-Controlled, Multiple-Ascending-Dose Investigation of the Oral Anti-Inflammatory Agent BT051 in Subjects With Moderately to Severely Active Ulcerative Colitis (UC)
Brief Title: An Investigation of Oral BT051 in Subjects With Moderately to Severely Active Ulcerative Colitis (UC)
Acronym: SCOUT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adiso Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT051-1-002
Record Dates: First submitted 2021-09-20; First posted 2021-10-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BT051 200 mg (Experimental): Participants will receive oral BT051 200 mg once daily for 28 days.
  Interventions: Drug: BT051 200 mg
- BT051 800 mg (Experimental): Participants will receive oral BT051 800 mg once daily for 28 days.
  Interventions: Drug: BT051 800 mg
- BT051 3200 mg (Experimental): Participants will receive oral BT051 3200 mg once daily for 28 days.
  Interventions: Drug: BT051 3200 mg
- Placebo (Placebo Comparator): Participants will receive oral Placebo to match BT051 once daily for 28 days.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: BT051 200 mg — Oral BT051 200 mg once daily for 28 days.
  Other Names: ADS051
  Arms: BT051 200 mg
Drug: BT051 800 mg — Oral BT051 800 mg once daily for 28 days.
  Other Names: ADS051
  Arms: BT051 800 mg
Drug: BT051 3200 mg — Oral BT051 3200 mg once daily for 28 days.
  Other Names: ADS051
  Arms: BT051 3200 mg
Drug: Matching Placebo — Placebo Matching BT051
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled study to assess the safety and tolerability of multiple ascending doses of BT051 in subjects with moderately to severely active ulcerative colitis. Subjects will be randomised using a 3 active:1 placebo ratio to 3 ascending dose cohorts of 8 subjects and will be dosed daily for 28 days. The 3 initial dose levels will be 200 mg, 800 mg and 3200 mg per day. Progression to the next cohort will be based on the safety and tolerability of the previous cohort.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, multiple-ascending-dose (MAD) study enrolling subjects with moderately to severely active UC. Subjects with prior exposure to biologic or JAK inhibitors will be limited to 30% of the total subject population; those who have failed 2 or more biologic therapies (i.e., biologic and JAK inhibitor, 2 biologics in the same class, or 2 biologics from different classes) will be limited to 20% of the total subject population. Subjects will be randomized to one of 3 doses of oral BT051 (200 mg, 800 mg, or 3200 mg) or placebo, in ascending dose groups based on the safety and tolerability of the previous cohort. Safety and tolerability will be assessed by a Safety Review Committee (SRC) after all subjects in each cohort have completed at least 14 days of treatment, before proceeding to the next higher dose cohort. The SRC may recommend that the next cohort proceed with a higher dose as planned, or the SRC may recommend additional subjects be dosed at the current, previous, or lower dose of study drug.

Each planned dose escalation cohort (Cohorts 1-3) will include 8 subjects randomized 3:1 to receive active drug or placebo. Starting with the lowest dose, each cohort of subjects will receive once daily oral BT051 or placebo for a period of 28 days. Follow-up visits will be performed at 7 and 30 days after the last dose.

ELIGIBILITY:
Inclusion Criteria

1. Provide written documentation of informed consent to participate in the study.
2. Male or female aged 18 to 75 years.
3. Subjects with a confirmed diagnosis of UC of at least 3 months' disease duration prior to Screening (diagnosis established by endoscopy and histology).
4. Moderately to severely active UC, defined as a Mayo Score ≥6 points with a rectal bleeding subscore ≥1 point, a stool frequency subscore ≥1 point, and moderate to severe disease on endoscopy (Mayo endoscopic subscore [MES] ≥2 points).
5. Subjects treated with stable doses (>4 weeks) of the following UC treatments prior to randomization: 6-mercaptopurine, azathioprine, sulfasalazine or 5-aminosalicylic acid. Subjects will need to maintain stable doses of these drugs for at least 4 weeks during study treatment and an additional 7 days of follow-up.
6. Subjects treated with oral corticosteroids will be eligible if the dose is ≤20 mg/day prednisone (≤9 mg/day budesonide) or equivalent. The corticosteroid therapy will have to be stable for at least 2 weeks prior to the Screening sigmoidoscopy, throughout study treatment and an additional 7 days of follow-up.
7. Colonoscopy within the past 1 year to exclude adenomas, dysplasia, and colon cancer for subjects with 1/3 of colon involved and 8 years of disease; those without a colonoscopy in the past year may use the Screening colonoscopy to confirm eligibility.
8. Female subjects must be surgically sterile, postmenopausal (i.e., no menses for at least 2 years or documented by follicle stimulating hormone), or if of child-bearing potential must have a negative pregnancy test and must be willing to use a highly effective form of contraceptive through 30 days after the last dose of study drug. The following are considered highly effective contraceptives: combined and progestogen-only hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal, injectable, implantable), intrauterine device/hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or abstinence. Abstinence should only be used as a contraceptive method if it is in line with the subject's usual and preferred lifestyle. Periodic abstinence (calendar, symptothermal, post ovulation methods) is not an acceptable method of contraception.
9. Male subjects must be surgically sterile, abstinent, agree to use an appropriate contraception method (i.e., condom), or have a female sexual partner who is surgically sterile, postmenopausal, or using a highly effective form of contraceptive as noted above through 30 days after the last dose of study drug. Abstinence should only be used as a contraceptive method if it is in line with the subject's usual and preferred lifestyle.

General Exclusion Criteria

1. Any clinically significant disease: renal, hepatic, neurological, cardiovascular, pulmonary, endocrinology, psychiatric, hematologic, urologic, or other acute or chronic disease that in the opinion of the Investigator would not make the subject a suitable candidate for this study.
2. Subjects with planned hospitalization or surgery during the course of the study.
3. Female subjects who have a positive pregnancy test, are breast feeding, or intend to become pregnant during the course of the study. Male subjects who intend female partner pregnancy during the course of the study.
4. Known hypersensitivity to any of the components of BT051 drug product including cyclosporine A and polyethylene glycol.
5. Relative to upper limit of normal (ULN):

   1. Serum bilirubin >1.5×
   2. Serum creatinine >1.5×
   3. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) >2.0×
6. International normalized ratio (INR) >1.5
7. Hemoglobin <8 g/dL
8. Cell counts (/μL):

   1. Platelets <100,000 or >800,000
   2. White blood cells <3500
   3. Absolute neutrophil count <1500
9. Systemic antibiotic, antiviral, or anti-fungal therapy within the 2 weeks prior to Screening.
10. Live or live-attenuated virus vaccination within the 2 weeks prior to randomization or planned vaccination during the study. Vaccination against SARS-CoV-2 using licensed vaccines will be permitted.
11. History of cancer within the past 5 years (permitted exceptions: subjects with excised basal cell carcinoma, squamous cell carcinoma of the skin, and cervical carcinoma in situ who have been treated and cured).
12. Drug, chemical, or alcohol dependency within the past 2 years as determined by the investigator.
13. A positive diagnostic tuberculosis (TB) test at screening (defined as a positive QuantiFERON test). In cases where the QuantiFERON test is indeterminate, the subject may have the test repeated once and if their second test is negative, they will be eligible. In the event a second test is also indeterminate, or QuantiFERON is unavailable, the investigator has the option to perform a purified protein derivative (PPD) skin test (PPD skin test may not be used if subject was previously vaccinated with bacille Calmette-Guerin [BCG]). If the PPD reaction is <5 mm, then the subject is eligible. If the reaction is ≥5 mm, or PPD testing is not done, the subject is not eligible.
14. Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) at Screening. If the initial test is positive but reflex testing (performed on the same sample) is negative, then the subject is eligible.
15. Inability to comply with study requirements.
16. Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment.
17. Subjects enrolled in another clinical trial assessing an investigational drug (or medical device) within 30 days or 5 half-lives (whichever is longer) prior to Screening (or within 60 days prior to Screening if investigational drug was a biologic).

    Gastrointestinal Exclusion Criteria
18. Fulminant colitis, toxic megacolon, or severe ulcerative colitis as defined: currently hospitalized for UC, fever, persistent tachycardia, or hemoglobin <8 g/dL.
19. Subject has any of the following conditions: primary sclerosing cholangitis, Crohn's disease, diverticulitis, bowel fistulas, history of colitis-associated colonic dysplasia, or active peptic ulcer disease.
20. Ulcerative colitis diagnosis limited to isolated proctitis.
21. Current ileostomy or colostomy.
22. Proctocolectomy or total colectomy.
23. Known symptomatic colonic stricture.
24. Current stool cultures or tests positive for an enteric infection, including parasitic infection and Clostridioides difficile toxin.
25. Short bowel syndrome requiring enteral or parenteral nutrition supplementation or total parenteral nutrition.
26. Diagnosis of microscopic or indeterminate colitis.
27. Bowel surgery within 3 months prior to randomization, or likely to need bowel surgery in next 4 months.
28. Any known history of listeria infection.
29. A current bacterial, parasitic, fungal, or viral infection (except blastocystis hominis).

    Prior Medication Exclusion Criteria
30. Prior biologic therapy:

    1. Adalimumab, infliximab, golimumab, etanercept, ustekinumab or certolizumab within the 60 days prior to Day 1.
    2. Vedolizumab within 120 days prior to Day 1.
31. Topical mesalamine or corticosteroid (i.e., enemas or suppositories) within the 14 days prior to Day 1.
32. Tofacitinib within the 30 days prior to Day 1.
33. Subjects treated with parenteral corticosteroids or calcineurin inhibitors cyclosporine, or tacrolimus within 4 weeks prior to randomization.
34. Regular use of other medications not mentioned above, including over-the-counter medications or supplements, that may impact the subject's UC or intestinal motility as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of BT051 based on the difference of proportions between treatment groups of subjects experiencing treatment-emergent adverse events (TEAEs) | Baseline to Day 58
  Proportion of subjects experiencing a TEAE will be summarized using the MedDRA system organ class and preferred term
Evaluate the safety and tolerability of BT051 based on the difference of proportions between treatment groups of subjects observed with a change from baseline in physical examinations, clinical laboratory tests, vital signs, and electrocardiograms (ECG) | Baseline to Day 58
  Proportion of subjects with a change from baseline from normal to abnormal in physical examinations, clinical laboratory tests, vital signs, and ECGs will be summarized

SECONDARY OUTCOMES:
Clinical response defined as a decrease in complete Mayo Score ≥3 points and ≥30% from baseline with a concomitant decrease in rectal bleeding subscore ≥1 point or absolute rectal bleeding subscore ≤1 point | Baseline to Day 28
  Proportion of subjects who achieve clinical response defined as a decrease in complete Mayo Score ≥3 points and ≥30% from baseline with a concomitant decrease in rectal bleeding subscore ≥1 point or absolute rectal bleeding subscore ≤1 point at Day 28
Clinical response defined as a decrease in complete Mayo Score ≥2 points and ≥30% from baseline with a concomitant decrease in rectal bleeding subscore ≥1 point or absolute rectal bleeding subscore ≤1 | Baseline to Day 28
  Proportion of subjects who achieve clinical response defined as a decrease in complete Mayo Score ≥2 points and ≥30% from baseline with a concomitant decrease in rectal bleeding subscore ≥1 point or absolute rectal bleeding subscore ≤1 point at Day 28
Remission defined as a complete Mayo Score ≤2 points with no subscore >1 point at Day 28 | Baseline to Day 28
  Proportion of subjects in clinical remission defined as a complete Mayo Score ≤2 points with no subscore >1 point at Day 28
Remission defined as a partial Mayo Score ≤2 points with no subscore >1 point at Days 14 and 28 | Baseline to Days 14 and 28
  Proportion of subjects in clinical remission defined as a partial Mayo Score ≤2 points with no subscore >1 point at Day 14 and Day 28
Remission according to the adapted Mayo Score without the physician's global assessment, defined as a stool frequency subscore ≤1 point, rectal bleeding subscore of 0, and endoscopic subscore ≤1 point | Baseline to Day 28
  Proportion of subjects in clinical remission according to the adapted Mayo Score without the physician's global assessment, defined as a stool frequency subscore ≤1 point, rectal bleeding subscore of 0, and endoscopic subscore ≤1 point
Change in Mayo endoscopic, stool frequency, and rectal bleeding subscores. | Baseline to Day 28
  Proportion of subjects with a change in Mayo endoscopic, stool frequency, and rectal bleeding subscores from baseline to Day 28
Change in stool frequency and rectal bleeding Mayo subscores | Baseline to Day 14
  Proportion of subjects with a change in stool frequency and rectal bleeding Mayo subscores from baseline to Day 14
Endoscopic remission defined as an Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score of 0 | Day 28
  Proportion of subjects who achieve endoscopic remission defined as an UCEIS score of 0 at Day 28
Endoscopic response defined as a decrease in UCEIS ≥2 points | Day 28
  Proportion of subjects who achieve endoscopic response defined as a decrease in UCEIS ≥2 points at Day 28.
Histologic remission defined as Geboes Score ≤2B.0 or Nancy Index = 0 | Day 28
  Proportion of subjects who achieve histologic remission (defined as Geboes Score ≤2B.0 or Nancy Index = 0) at Day 28
Change in Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score | Baseline to Day 28
  Difference between treatment groups of mean change in UCEIS score from baseline to Day 28.
  The UCEIS consists of the following 3 descriptors and is calculated as a simple sum: erosions and ulcers (scored 0-3), bleeding (scored 0-3) and vascular pattern (scored 0-2). Calculated scores range from 0 to 8 with higher scores indicating more severe disease.
Change in Robarts histopathology index (RHI) score | Baseline to Day 28
  Difference between treatment groups of mean change in Robarts histopathology index (RHI) score from baseline to Day 28.
  The RHI score ranges from 0 (no disease activity) to 33 (severe disease activity) based on the evaluation of 4 main parameters: chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in the epithelium, and erosion and ulceration.
Change in UC-100 score | Baseline to Day 28
  Difference between treatment groups of mean change in UC-100 score from baseline to Day 28.
  The UC-100 is a composite disease activity index consisting of clinical, endoscopic, and histological findings. The UC-100 will be calculated by adding the weighted Mayo stool frequency and endoscopy subscores, and RHI score as follows:
  UC-100 Score = 1 + (16 × stool frequency) + (6 × MES) + (RHI score)
  The total UC-100 score ranges from 1 to 100, with higher scores representing more severe disease activity.

OTHER OUTCOMES:
Maximum observed concentration (Cmax) in whole blood | Baseline to Day 28
  Difference between treatment groups of mean Cmax of BT051 and BT070 in whole blood
Time to maximum observed concentration (Tmax) in whole blood | Baseline to Day 28
  Difference between treatment groups of mean Tmax of BT051 and BT070 in whole blood
Area Under the Concentration-Time Curve (AUC) in whole blood | Baseline to Day 28
  Difference between treatment groups of mean AUC of BT051 and BT070 in whole blood
Total Body Clearance (CL) in whole blood | Baseline to Day 28
  Difference between treatment groups of mean CL of BT051 and BT070 in whole blood
BT051 and BT070 concentrations in stool, colonic tissue, and urine | Baseline to Day 58
  Difference of means between treatment groups in concentrations of BT051 and BT070 in stool, colonic tissue, and urine.

CONTACTS AND LOCATIONS:
Overall Officials: Renu Gupta, MD, Study Director — Adiso Therapeutics, Inc.
Locations (6):
- United States (2):
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - I.H.S. Health, LLC, Kissimmee, Florida
- Research Institute of Clinical Medicine Todua Clinic, Tbilisi, Georgia
- Republican Clinical Hospital - Timofei Mosneaga, Chisinau, Moldova
- Poland (2):
  - WIP Warsaw IBD Point, Warsaw
  - PlanetMed Gastroenterology, Wroclaw

REFERENCES:
- [Derived] Allegretti JR, Cheifetz AS, Dulai PS, Stevens AC, Chapas-Reed J, Chesnel L, Dixit B, Farquhar R, Ghahramani P, Miller BW, Murphy CK, Quintas M, Tanase R, Telia T, Wozniak-Stolarska B, Gupta R. Safety, Pharmacokinetics, and Clinical Efficacy of ADS051, a Neutrophil Modulator, in Ulcerative Colitis: Results of a Randomized Phase 1b Trial. Am J Gastroenterol. 2024 Dec 31;120(7):1624-1635. doi: 10.14309/ajg.0000000000003269. PMID 39787364